CLINICAL TRIAL: NCT00285623
Title: An Non-interventional, Prospective, Non-controlled Study of the Use of TachoSil in Supportive Treatment in Surgery for Improvement of Haemostasis Where Standard Techniques Are Insufficient.
Brief Title: Observational Cohort Study of TachoSil (TC-018-IN)
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Clinical Trial Operations
Other Study IDs: TC-018-IN
Record Dates: First submitted 2005-12-21; First posted 2006-02-02 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2009-07

CONDITIONS: Blood Loss, Surgical
Keywords: Collection of all thromboembolic events,; immunological events and drug interactions leading to thromboembolic events or major; bleeding after exposure to TachoSil®.
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Fibrinogen; Thrombin; TachoSil

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fibrinogen (human) + thrombin (human) (TachoSil) — treatment in surgery for improvement of haemostasis where standard techniques are insufficient

SUMMARY:
The purpose of this study is to collect information, after exposure to TachoSil ®, of all thromboembolic events, immunological events and drug interactions leading to thromboembolic events or major bleeding. In addition, pharmacoeconomic data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* All subjects, treated with TachoSil ® by the participating physicians, will be registered with a set of basic data from their already existing data (i.e. no additional diagnostic procedures will be performed).
* Subjects who will provide their written informed consent to use existing data, allow direct access to data and data processing.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients exposed to TachoSil® of all thromboembolic events, immunological events and drug interactions leading to thromboembolic events or major bleeding.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2005-12; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquarters
Locations (1):
- Nycomed, Roskilde, Denmark

REFERENCES:
- [Derived] Birth M, Figueras J, Bernardini S, Troen T, Gunther K, Mirza D, Mortensen FV. Collagen fleece-bound fibrin sealant is not associated with an increased risk of thromboembolic events or major bleeding after its use for haemostasis in surgery: a prospective multicentre surveillance study. Patient Saf Surg. 2009 Jun 22;3(1):13. doi: 10.1186/1754-9493-3-13. PMID 19545437